CLINICAL TRIAL: NCT02909257
Title: Minimum Effective Concentration of Bupivacaine for Motor-Sparing Femoral Nerve Block
Brief Title: Motor-Sparing Femoral Nerve Block Dose
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inadequate methodology to determine primary outcome
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, MD, Attending Anesthesiologist, Clinical Instructor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OAIC 823/16
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee; Knee Injuries
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- same dose (Experimental): patient is exposed to the same previously successful dose
  Interventions: Drug: Same Bupivacaine Concentration
- lower dose (Experimental): patient is exposed to a lower concentration dose
  Interventions: Drug: Lower Bupivacaine Concentration

INTERVENTIONS:
Drug: Same Bupivacaine Concentration — patient is exposed to the same concentration than previously successful one
  Arms: same dose
Drug: Lower Bupivacaine Concentration — patient is exposed to a lower concentration than previously successful one
  Arms: lower dose

SUMMARY:
Femoral nerve blocks are commonly used to provide pain control for total knee replacement, anterior cruciate ligament (ACL) reconstruction. Commonly employed local anesthetic concentrations result in motor block of the quadriceps and constitute an inherent risk factor for patient fall.

The aim of this study is to determine the minimum effective concentration of bupivacaine in 90 % of patients (MEC90) required for a motor-sparing, successful sensory block of the femoral nerve.

DETAILED DESCRIPTION:
With the approval of Ethics Committee of the University of Chile Clinical Hospital, approximately 60 patients undergoing ACL repair or TKR will be recruited. All blocks will be conducted preoperatively in an induction room.Dose assignation will be done using an up-and-down sequential method, where the dose of each subsequent patient depends on the response of the previous patient, called the Biased Coin Design.

The assignment of each subsequent concentration will be based on the response of the previous patient.As soon as we recruit 45 patients with random dose assignment, we will terminate the enrollment procedure.

The injectate will be prepared and administered by a research assistant using syringes connected to the block needle. The operator and the patient will be blinded to the concentration injected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets≤ 100, International Normalized Ratio≥ 1.4 or partial prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to LA
* Pregnancy
* Prior surgery in the inguinal region
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Minimum Bupivacaine Analgesic concentration preserving quadriceps strength analgesia | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: DE QH TRAN, MD, FRCPC, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Hospital Clinico Universidad de Chile, Santiago, Metropolitan, Chile

REFERENCES:
- [Result] Biboulet P, Morau D, Aubas P, Bringuier-Branchereau S, Capdevila X. Postoperative analgesia after total-hip arthroplasty: Comparison of intravenous patient-controlled analgesia with morphine and single injection of femoral nerve or psoas compartment block. a prospective, randomized, double-blind study. Reg Anesth Pain Med. 2004 Mar-Apr;29(2):102-9. doi: 10.1016/j.rapm.2003.11.006. PMID 15029544
- [Result] Dauri M, Sidiropoulou T, Fabbi E, Giannelli M, Faria S, Mariani P, Sabato AF. Efficacy of continuous femoral nerve block with stimulating catheters versus nonstimulating catheters for anterior cruciate ligament reconstruction. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):282-7. doi: 10.1016/j.rapm.2006.06.249. PMID 17720111
- [Result] Schiferer A, Gore C, Gorove L, Lang T, Steinlechner B, Zimpfer M, Kober A. A randomized controlled trial of femoral nerve blockade administered preclinically for pain relief in femoral trauma. Anesth Analg. 2007 Dec;105(6):1852-4, table of contents. doi: 10.1213/01.ane.0000287676.39323.9e. PMID 18042893
- [Result] Johnson RL, Kopp SL, Hebl JR, Erwin PJ, Mantilla CB. Falls and major orthopaedic surgery with peripheral nerve blockade: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):518-28. doi: 10.1093/bja/aet013. Epub 2013 Feb 24. PMID 23440367
- [Result] Casati A, Fanelli G, Beccaria P, Magistris L, Albertin A, Torri G. The effects of single or multiple injections on the volume of 0.5% ropivacaine required for femoral nerve blockade. Anesth Analg. 2001 Jul;93(1):183-6. doi: 10.1097/00000539-200107000-00036. PMID 11429362
- [Result] Jaeger P, Koscielniak-Nielsen ZJ, Hilsted KL, Fabritius ML, Dahl JB. Adductor Canal Block With 10 mL Versus 30 mL Local Anesthetics and Quadriceps Strength: A Paired, Blinded, Randomized Study in Healthy Volunteers. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):553-8. doi: 10.1097/AAP.0000000000000298. PMID 26237001
- [Result] Lu YM, Lin JH, Hsiao SF, Liu MF, Chen SM, Lue YJ. The relative and absolute reliability of leg muscle strength testing by a handheld dynamometer. J Strength Cond Res. 2011 Apr;25(4):1065-71. doi: 10.1519/JSC.0b013e3181d650a6. PMID 20838248
- [Result] Lu TW, Hsu HC, Chang LY, Chen HL. Enhancing the examiner's resisting force improves the reliability of manual muscle strength measurements: comparison of a new device with hand-held dynamometry. J Rehabil Med. 2007 Nov;39(9):679-84. doi: 10.2340/16501977-0107. PMID 17999004
- [Result] Tran DQ, Dugani S, Dyachenko A, Correa JA, Finlayson RJ. Minimum effective volume of lidocaine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):190-4. doi: 10.1097/AAP.0b013e31820d4266. PMID 21270721
- [Result] Stylianou M, Flournoy N. Dose finding using the biased coin up-and-down design and isotonic regression. Biometrics. 2002 Mar;58(1):171-7. doi: 10.1111/j.0006-341x.2002.00171.x. PMID 11890313